CLINICAL TRIAL: NCT01806194
Title: Empowering Rural African American Women and Communities to Improve Diabetes Outcomes
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Doyle M. Cummings, Professor of Family Medicine, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 212196
Record Dates: First submitted 2012-12-05; First posted 2013-03-07 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational control arm (Active Comparator): Control group receives 16 mailings of diabetes educational materials but no regular contact with community health workers
  Interventions: Behavioral: Educational Control Arm
- Lifestyle counseling (Experimental): Small changes behavioral counseling and social support, delivered in 16 sessions by community health workers.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Small changes behavioral counseling and social support, delivered in 16 sessions by community health workers
  Arms: Lifestyle counseling
Behavioral: Educational Control Arm — 16 mailings of diabetes educational materials but no regular contact with community health workers
  Arms: Educational control arm

SUMMARY:
The EMPOWER diabetes program is a year-long, community-based program designed to enhance diabetes management in rural African American women with uncontrolled diabetes. The treatment is delivered by community peers and follows a relative Small Changes approach.

DETAILED DESCRIPTION:
East Carolina University, along with established community partners, is implementing a community-based and culturally-tailored intervention to reduce diabetes disparities in 200 rural African American women with uncontrolled diabetes using our unique behaviorally-centered small changes approach to diabetes self-management, delivered by community health workers. The focus is on moderation and patient-selected small changes in eating, activity, and care management that decrease feelings of deprivation and failure and increase feelings of confidence and success. The intervention is specifically tailored to overcome psychosocial and environmental barriers to behavioral change through a strong focus on emotional, cultural, and social factors related to eating, activity, and medications. Objectives for the proposed project are to: 1) implement and evaluate the effectiveness of this tailored small changes intervention; 2) examine the impact of this approach on psychological mediators of behavioral choices in diabetes; 3) implement and evaluate public policy and built environment advocacy strategies; and 4) build, sustain, and disseminate a business-sustainable care model. The study will be a randomized prospective trial comparing the small changes intervention, delivered in 16 sessions by community health workers, to a control group receiving 16 mailings of diabetes educational materials. We hypothesize that there will be a greater improvement in behavioral choices and glycemic control in the intervention group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* African American female,
* age 19 - 75yr.,
* with Type 2 diabetes mellitus and
* living in or near Bertie, Edgecombe, and Pitt counties in eastern NC

Exclusion Criteria:

-

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | 6 months
  Glycosylated hemoglobin
Change in Hemoglobin A1c | 12 Months
  Glycosylated hemoglobin

SECONDARY OUTCOMES:
Change in Weight | 6 Months
  Body weight
Change in Weight | 12 Months
  Body Weight

OTHER OUTCOMES:
Blood pressure | 6 months
  Blood pressure
Blood Pressure | 12 Months
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Doyle M. Cummings, Pharm.D., Principal Investigator — East Carolina University; Lesley Lutes, Ph.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Cummings DM, Lutes LD, Littlewood K, Dinatale E, Hambidge B, Schulman K. EMPOWER: a randomized trial using community health workers to deliver a lifestyle intervention program in African American women with Type 2 diabetes: design, rationale, and baseline characteristics. Contemp Clin Trials. 2013 Sep;36(1):147-53. doi: 10.1016/j.cct.2013.06.006. Epub 2013 Jun 19. PMID 23792133
- [Background] Cummings DM, Lutes L, Littlewood K, DiNatale E, Hambidge B, Schulman K, Morisky DE. Regimen-Related Distress, Medication Adherence, and Glycemic Control in Rural African American Women With Type 2 Diabetes Mellitus. Ann Pharmacother. 2014 Aug;48(8):970-977. doi: 10.1177/1060028014536532. Epub 2014 Jun 5. PMID 24904183
- [Derived] Lutes LD, Cummings DM, Littlewood K, Dinatale E, Hambidge B. A Community Health Worker-Delivered Intervention in African American Women with Type 2 Diabetes: A 12-Month Randomized Trial. Obesity (Silver Spring). 2017 Aug;25(8):1329-1335. doi: 10.1002/oby.21883. Epub 2017 Jun 29. PMID 28660719